CLINICAL TRIAL: NCT06644820
Title: Clinical Characteristics and Outcome of Patients Xith Spontaneous Pneumothorax
Status: Recruiting | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Yassmin Mehana Aboelfadel, resident-chest department sohag university hospital, Sohag University
Other Study IDs: Soh-Med-24-09-14MS
Record Dates: First submitted 2024-10-08; First posted 2024-10-16 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2024-10

CONDITIONS: Spontaneous Pneumothorax
MeSH Terms: conditions — Pneumothorax | interventions — Diagnostic Imaging

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Primary spontaneous pneumothorax: Primary spontaneous pneumothorax (PSP) occur in the absence of underlying lung disease. Primary spontaneous pneumothorax is more common in men and in younger patients and associated with smoking.
  Interventions: Diagnostic Test: radiology
- Secondary spontaneous pneumothorax: Secondary spontaneous pneumothorax (SSP) occur in the presence of underlying lung disease, most commonly chronic obstructive pulmonary disease, cystic fibrosis, pneumocystis pneumonia, lung cancer, and interstitial lung diseases (ILDs) in older adults.
  Interventions: Diagnostic Test: radiology

INTERVENTIONS:
Diagnostic Test: radiology — Chest x ray posteroanterior view and lateral view.
  CT. chest without contrast:
  To assess the underlying lung pathology e.g. multiple bullae, interstitial lung disease (ILD) , cavitating lesions or nodules.

SUMMARY:
Pneumothorax occurs when air accumulates between the visceral and parietal pleura, and canbe defined as spontaneous, iatrogenic or traumatic. Spontaneous pneumothorax further classified as primary or secondary. Primary spontaneous pneumothorax (PSP) occur in the absence of underlying lung disease. Primary spontaneous pneumothorax is more common in men and in younger patients and associated with smoking. Secondary spontaneous pneumothorax (SSP) occur in the presence of underlying lung disease, most commonly chronic obstructive pulmonary disease, cystic fibrosis, pneumocystis pneumonia, lung cancer,and interstitial lung diseases (ILDs) in older adults.

ELIGIBILITY:
Inclusion Criteria:

* The study will include patients ≥18 years old with spontaneous pneumothorax admitted at Sohag University Hospital

Exclusion Criteria:

* Patients with traumatic or iatrogenic pneumothorax.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will include patients ≥18 years old with spontaneous pneumothorax admitted at Sohag University Hospital
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-10-30 (Estimated); Study Completion 2025-10-30 (Estimated)

PRIMARY OUTCOMES:
Duration of hospital stay | 1 year
  hospitalization time of patients with spontanous pneumothorax from addmission to discharge from hospital

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag university Hospital, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Graham BL, Steenbruggen I, Miller MR, Barjaktarevic IZ, Cooper BG, Hall GL, Hallstrand TS, Kaminsky DA, McCarthy K, McCormack MC, Oropez CE, Rosenfeld M, Stanojevic S, Swanney MP, Thompson BR. Standardization of Spirometry 2019 Update. An Official American Thoracic Society and European Respiratory Society Technical Statement. Am J Respir Crit Care Med. 2019 Oct 15;200(8):e70-e88. doi: 10.1164/rccm.201908-1590ST. PMID 31613151
- [Background] Hilliard NJ, Marciniak SJ, Babar JL, Balan A. Evaluation of secondary spontaneous pneumothorax with multidetector CT. Clin Radiol. 2013 May;68(5):521-8. doi: 10.1016/j.crad.2012.10.008. Epub 2012 Dec 5. PMID 23218593
- [Background] Khusial RJ, Honkoop PJ, van der Meer V, Snoeck-Stroband JB, Sont JK. Validation of online Asthma Control Questionnaire and Asthma Quality of Life Questionnaire. ERJ Open Res. 2020 Jan 27;6(1):00289-2019. doi: 10.1183/23120541.00289-2019. eCollection 2020 Jan. PMID 32010723
- [Background] Noh TJ, Lee CH, Kang YA, Kwon SY, Yoon HI, Kim TJ, Lee KW, Lee JH, Lee CT. Chest computed tomography (CT) immediately after CT-guided transthoracic needle aspiration biopsy as a predictor of overt pneumothorax. Korean J Intern Med. 2009 Dec;24(4):343-9. doi: 10.3904/kjim.2009.24.4.343. Epub 2009 Nov 27. PMID 19949733